CLINICAL TRIAL: NCT02977845
Title: Effect of Qigong on the Symptom Clusters of Dyspnea, Fatigue, and Anxiety.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nam Dinh University of Nursing (Other)
Collaborators: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, VU VAN DAU, Senior lecturer, Nam Dinh University of Nursing
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: NamDUN
Record Dates: First submitted 2016-11-26; First posted 2016-11-30 (Estimated); Last update posted 2018-06-28 (Actual); Status verified 2018-06

CONDITIONS: Lung Cancer, Nonsmall Cell; Lung Cancer Non-Small Cell Stage 0; Lung Cancer, Nonsmall Cell, Stage I; Lung Cancer Non-Small Cell Stage II; Lung Cancer, Limited Stage Small Cell
Keywords: dypsnea; fatigue; anxiety; Qigong; Lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Fatigue; Anxiety Disorders | interventions — Qigong

STUDY DESIGN:
Intervention Model Description: The design of this study was a randomized controlled trial (RCT) with two parallel groups in a 1:1 allocation ratio, allocation concealment, and assessor blinding.
Who Masked: Outcomes Assessor
Masking Description: In the current study, based on nature of the intervention, blinding was not feasible with researcher, statistician, Qigong master who were responsible for recruitment of subject, randomization, deliver the intervention. However, the investigators who collect the outcome information were blinded to the allocation sequence.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Primary aim (Experimental): The primary aim of this study is to assess the effect of Qigong on managing dyspnea, fatigue, and anxiety (as a cluster) in lung cancer patients.
  Interventions: Behavioral: Qigong
- Secondary aim (Experimental): The secondary aim of this study is exploring the effect of Qigong on cough which is another common symptom linked with dyspnea, fatigue, and anxiety as a cluster, and QOL in lung cancer patients.
  Interventions: Behavioral: Qigong

INTERVENTIONS:
Behavioral: Qigong — Qigong has long been regarded as a form of "mind-body" intervention in Traditional Chinese Medicine (TCM), which simultaneously exercises the "mind" and the "body" for treating many chronic diseases and promoting wellness. About a hundred million people are currently practicing Qigong in China. Qigong is now regarded as a form of self-practise mind-body exercise and recently relevant to sports activity, which is officially known as "Health Qigong". It is different from "Medical Qigong" which involves a TCM practitioner to emit "Qi" to heal the patients.
  Other Names: Chi Kung

SUMMARY:
Effects of Qigong on symptom clusters of dyspnea, fatigue, and anxiety in Vietnamese lung cancer patients: A randomized control trial

DETAILED DESCRIPTION:
Background: Patients with lung cancer experience a variety of symptoms. The number of symptoms ranged from 7.8 to 13.2, and most of them were at a moderate level of severity. Dyspnea, fatigue, and anxiety arose as the most problematic symptoms of lung cancer. Non-pharmacological approaches to manage of symptom among lung cancer patients showed either no or mild effects. Qigong is hypothesized to alleviate these adverse outcomes; however, all trial analyzed on a single symptom, and not lung cancer patients, and there have not been many well-designed randomized control trials. The objectives of this study are following: 1) to assess the effect of Qigong on managing dypsnea, fatigue, and anxiety (as a cluster) in lung cancer patients; 2) to explore the effect of Qigong on cough another common symptom linked with dyspnea, fatigue as a cluster and quality of life (QOL) in lung cancer patients.

Methods: 156 subjects with lung cancer (stage I - IV) will be randomized to either the Qigong group or the wait-list control group. Participants in the Qigong group will conduct Qigong practice 5 times per week for 6 weeks, and participants in the control group will receive usual care. The primary outcome (dypsnea, fatigue, and anxiety), secondary outcomes (cough and QOL) will be assessed at baseline, post-intervention, and post 6-weeks of follow-up.

Discussion: This study will be the first randomized trial to investigate the effectiveness of Qigong for management symptom cluster in lung cancer patients. The finding of this study will help to establish the optimal approach for the care of lung cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed of lung cancer [Non-small cell lung cancer (NSCLC) or Small cell lung cancer (SCLC)];
* Patients with Stage I - III NSCLC or SCLC and have completed treatment with chemotherapy and/or radiotherapy for a minimum of 4 weeks prior to commencing the study;
* Medically fit to participate in general well-being and activities of daily life, as two or smaller on a 0 - to 5-point numeric rating scale at the time of recruitment, as determined by The Eastern Cooperative Oncology Group (ECOG) score;
* With no evidence of recurrence or occurrence of other cancers; and
* Patients report all three symptoms (dyspnea, fatigue, and anxiety) in the previous week and ranked the severity of at least two of the three symptoms as 3 or more on a 0 - to 10-point numeric rating scale at the time of recruitment, as determined by dyspnea, fatigue, and anxiety intensity rating scale

Exclusion Criteria:

* Clinically diagnosed with major psychiatric illness;
* Presenting with criteria associated with risk during physical activity: severe cachexia; frequent dizziness; bone pain; or severe nausea;
* Having had past or current regular experience with mind-body practices that blend movement with meditative practices, such as Yoga, Tai Chi, or Qigong;
* Life expectancy of < 6 months (as determined by their physicians).
* Visual problems or deafness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-06-22 (Actual)

PRIMARY OUTCOMES:
A cluster symptom of dyspnea, fatigue, and anxiety in lung cancer patients. | 12 weeks
  * Dyspnea is described as "an uncomfortable awareness of breathing" (DiSalvo, Joyce, Tyson, Culkin, & Mackay, 2008). Cancer Dyspnoea Scale will be used to measure dypsnea in this study.
  * Fatigue is defined as "a subjective feeling of tiredness, weakness or lack of energy" (Radbruch et al., 2008). Functional Assessment of Cancer Therapy-Fatigue (FACT-F) (Yellen et al., 1997) will be used to measure fatigue in this study.
  * Anxiety is defined as "The apprehensive anticipation of future danger or misfortune accompanied by a feeling of dysphoria or somatic symptoms of tension" (American Psychiatric Association, 2005). The Anxiety subscale of the Depression, Anxiety, and Stress Scale 21 (DASS-21) (Sharp et al., 2013) will be used to measure anxiety in this study.

SECONDARY OUTCOMES:
Cough | 12 weeks
  Cough is "a forced expulsive manoeuvre, usually against a closed glottis and which is associated with a characteristic sound" (McGarvey & Morice, 2006; Pavord & Chung, 2008). Manchester Cough in Lung Cancer Scale (MCLCS) (Molassiotis et al., 2012) will be used to measure cough in this study.
Quality of Life | 12 weeks
  The World Health Organization (WHO) defined health as "a state of complete physical, mental and social well-being and not merely the absence of disease or infirmity". European Organization for Research and Treatment of Cancer -Quality of life questionnaire - Core and Lung module (Fayers et al., 2012) will be used to measure quality of life in this study.

CONTACTS AND LOCATIONS:
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided
Later

REFERENCES:
- [Derived] Molassiotis A, Vu DV, Ching SSY. The Effectiveness of Qigong in Managing a Cluster of Symptoms (Breathlessness-Fatigue-Anxiety) in Patients with Lung Cancer: A Randomized Controlled Trial. Integr Cancer Ther. 2021 Jan-Dec;20:15347354211008253. doi: 10.1177/15347354211008253. PMID 33847150